CLINICAL TRIAL: NCT02480244
Title: Translating Obesity and Diabetes Prevention Into the Worksite for Immigrant Populations
Brief Title: PASOS: Improving the Health of Immigrant Workers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Davis (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 575576; R18DK096429 (NIH)
Record Dates: First submitted 2015-06-09; First posted 2015-06-24 (Estimated); Last update posted 2020-08-07 (Actual); Status verified 2020-08

CONDITIONS: Overweight and Obesity; Diabetes
MeSH Terms: conditions — Overweight; Obesity; Diabetes Mellitus | interventions — Behavior Therapy; Diet

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Behavioral intervention (Experimental): Behavioral intervention consisting of 12 educational sessions promoting healthy diet and increased physical activity
  Interventions: Behavioral: Behavioral Intervention
- Control (Active Comparator): Control arm receives no health-related behavioral intervention
  Interventions: Other: Control

INTERVENTIONS:
Behavioral: Behavioral Intervention — Intervention participants attend up to 12 educational sessions teaching them about diabetes, and modifiable lifestyle factors (behaviors) to reduce the risk of diabetes by controlling weight. Sessions are conducted by Promotoras using culturally sensitive and appropriate materials and themes. Group activities and support are also emphasized. The control participants like the intervention were measured and interviewed before and again after the intervention sessions, but received no educational instruction or materials.
  Other Names: Healthy Lifestyle intervention; Diet and Physical Activity intervention
  Arms: Behavioral intervention
Other: Control — Control arm receives no health-related behavioral intervention
  Arms: Control

SUMMARY:
This is a cluster randomized trial (CRT) to assess the effectiveness of a culturally appropriate behavioral intervention to reduce obesity levels and ultimately the risk of developing diabetes type II in immigrant Latino farm workers. Randomization is at the farm ranch level. Individuals at intervention ranches will receive a multi-week curriculum at the work-site on diabetes, diet and physical activity and optional supplemental sessions in the evening and weekends. The investigators will adopt the intent-to-treat principle for the primary analysis. Individuals on control ranches will receive no health educational instruction. The primary outcome is BMI. The investigators hypothesize that intervention ranches will achieve significant improvement in obesity and diabetes risk factors as compared to control ranches.

ELIGIBILITY:
Inclusion Criteria:

* Work at Reiter Brothers Inc. (RBI), a partner, or affiliate company
* Able to speak and understand Spanish
* Willing to attend weekly sessions for length of intervention
* Plan to stay in the area for the next three months

Exclusion Criteria:

* Workers without Spanish language comprehension
* Pregnant women and those planning a pregnancy within six months
* Women who are breastfeeding, unless discontinuing breastfeeding within one month
* Individuals who, without health care provider approval, are: unable to undertake moderate physical exercise, taking medicine for high blood pressure or heart conditions, have bone or joint problems, lose consciousness or fall due to dizziness, or have developed chest pain within the last month
* Individuals taking medications that affect weight
* Individuals with therapeutic diets
* Diabetic status determined by health care professional after HbA1c testing result is >6.5%
* If spouse / cohabitant is already in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 554 (Actual)
Dates: Start 2015-07 (Actual); Primary Completion 2018-10-02 (Actual); Study Completion 2018-10-02 (Actual)

PRIMARY OUTCOMES:
Change in BMI | Measured at baseline prior to the intervention; immediately following the intervention (12 weeks after first assessment) and again at 6 months, 1 year, and 1.5 years post-intervention.
  Weight and height will be assessed at each data collection point and concurrently for control and intervention participants on matched ranches.

SECONDARY OUTCOMES:
Change in waist circumference | Measured at baseline prior to the intervention; immediately following the intervention (12 weeks after first assessment) and again at 6 months, 1 year, and 1.5 years post-intervention.
  Waist circumference will be assessed concurrently for control and intervention participants on matched ranches using a standard protocol.
Change in hemoglobin A1c (HbA1c) | Measured at baseline prior to the intervention; immediately following the intervention (12 weeks after first assessment) and again at 1 year post-intervention.
  HbA1c will be assessed concurrently for control and intervention participants on matched ranches using a standard protocol.
Change in cholesterol | Measured at baseline prior to the intervention; immediately following the intervention (12 weeks after first assessment) and again at 1 year post-intervention.
  Cholesterol will be assessed concurrently for control and intervention participants on matched ranches using a standard protocol.
Change in behavior and lifestyle factors | Measured at baseline prior to the intervention; immediately following the intervention (12 weeks after first assessment) and again at 1 year post-intervention.
  Change in behavior and lifestyle factors will be assessed concurrently for control and intervention participants on matched ranches using a questionnaire comprised of validated measures.
Cost analysis | Quarterly beginning a year prior to implementation of the intervention and concluding 1.5 years post-intervention.
  Assessment of intervention's impact on employer costs.
Change in blood pressure | Measured at baseline prior to the intervention; immediately following the intervention (12 weeks after first assessment) and again at 6 months, 1 year, and 1.5 years post-intervention.
  Change in blood pressure will be assessed concurrently for control and intervention participants on matched ranches using a standard protocol.

CONTACTS AND LOCATIONS:
Overall Officials: Marc Schenker, MD, MPH, Principal Investigator — University of California, Davis
Locations (1):
- Reiter Brothers Inc., Oxnard, California, United States

REFERENCES:
- [Derived] Borelli MR, Riden HE, Bang H, Schenker MB. Protocol for a cluster randomized controlled trial to study the effectiveness of an obesity and diabetes intervention (PASOS) in an immigrant farmworker population. BMC Public Health. 2018 Jul 9;18(1):849. doi: 10.1186/s12889-018-5560-0. PMID 29986676